CLINICAL TRIAL: NCT03938480
Title: Duration Threstholds of Intraoperative Hypotension for Postoperative Major Adverse Events
Brief Title: Duration Threstholds of Intraoperative Hypotension
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Yan Zhou, MD, Principal Investigator, Peking University First Hospital
Other Study IDs: DTIH
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intraoperative hypotension is common in non cardiac surgery. longer duration of intraoperative hypotension is related with postoperative morbidity and mortality. however, with the change of hypotension criteria, the duration threshold also change. the relationship of different hypotension criteria and its duration is unclear. This study is to explore the their relationship.

DETAILED DESCRIPTION:
Intraoperative hypotension is common in non cardiac surgery. longer duration of intraoperative hypotension is related with postoperative morbidity and mortality. however, with the change of hypotension criteria, the duration threshold also change. the relationship of different hypotension criteria and its duration is unclear. This study is to explore the relationship between continous difference mean blood pressure criteria and its duration thresholds for postoperative major adverse events, which include acute cardiac infarction, heart failure, cardiac death, stroke and acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

adults underwent elective non-cardiac surgery

Exclusion Criteria:

cardiac surgeries; kidney surgeries; obstetric surgeries; local infiltration anesthesia; surgeries without arterial pressure monitoring; perioperative data missing; patients with more than one operation within a year

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The analysis set of this study was adults (age ≥ 18 years old) who underwent elective non-cardiac surgery from January 1, 2012, to December 31, 2017.
Sampling Method: Non-Probability Sample
Enrollment: 37000 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-22 (Actual)

PRIMARY OUTCOMES:
major adverse events | 30 days postoperatively in hospital
  including acute cardiac infarction, heart failure, cardiac death, stroke, kidney injury

CONTACTS AND LOCATIONS:
Locations (1):
- PKU 1st hospital, Beijing, Beijing Municipality, China